CLINICAL TRIAL: NCT07073508
Title: The Validity of the Evaluation of Renal Artery Duplex in Critically Ill Acute Kidney Injury Patients
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mahmoud rabie, Assistant Lecturer of Anesthesiology, Intensive Care and Pain Management, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Other Study IDs: FMASU MD51/2024
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Validity; Renal Artery Duplex; Critically Ill Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients diagnosed with acute kidney injury (AKI).
  Interventions: Other: Renal Artery Duplex

INTERVENTIONS:
Other: Renal Artery Duplex — Renal artery duplex will be performed to all patients in terms of renal resistivity index (RRI).

SUMMARY:
This study aims to assess the clinical relevance of renal artery duplex ultrasound in critically ill patients with acute kidney injury (AKI) in terms of the renal resistive index (RRI).

DETAILED DESCRIPTION:
Diagnosis of acute kidney injury (AKI) is based on rising creatinine as late phenomenon. Intrarenal vasoconstriction occurs earlier, so measuring flow resistance in the renal circulation, renal resistive index (RRI), could become part of vital organ function assessment using Doppler ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients age >18 years.
* Both sexes.
* Patients within 24 hours after intensive care unit (ICU) admission.

Exclusion Criteria:

* Patients presented with poor abdominal echogenicity.
* Chronic kidney disease, especially with estimated creatinine clearance less than 30 ml/min/1.73m.
* Patients with dialysis dependency.
* Patients with renal transplantation.
* Patients with known renal artery stenosis.
* If there is a pregnancy.
* Patients with any congenital kidney diseases as mono-kidney, anatomic kidney abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred patients admitted to the intensive care unit (ICU), all the studied populations will be diagnosed to have AKI, with no past medical history of chronic renal disease.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Renal resistivity index (RRI) | 1 week post-procedure
  The renal resistivity index (RRI) will be assessed in patients with acute kidney injury (AKI) who require intensive care unit (ICU) admission within 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.